CLINICAL TRIAL: NCT05774522
Title: Study of Anatomo-functional Correlation of the Upper Airways
Acronym: P3E
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: APHP220939; 2022-A01754-39 (Other: EUDRACT)
Record Dates: First submitted 2023-02-22; First posted 2023-03-17 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Sleep Apnea Syndromes
Keywords: sleep apnea syndrome; upper airway; pCrit; acoustic pharyngometry; upper airway ultrasound
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Suspicion of sleep apnea syndrome (Experimental): All patients, consulting Bichat sleep center for suspected sleep apnea syndrome
  Interventions: Other: Measurement of pharyngeal critical airway closing pressure; Other: Acoustic pharyngometry; Other: Upper airway ultrasound

INTERVENTIONS:
Other: Measurement of pharyngeal critical airway closing pressure — The Pcrit will be measured on an automatic controlled device specially designed by the engineers of the inserm neophen team capable of varying the pressures from +4 to -20 centimeters of water, by a nasal mask whose pressures are connected to a pneumotachograph. The measurements will be performed in supine position.
  Other Names: pCrit
Other: Acoustic pharyngometry — Acoustic pharyngometry is an non-invasive technique consisting of the propagation of an acoustic wave from the lips to the larynx providing information on the lengths, cross-sectional areas and volumes of the air spaces.
Other: Upper airway ultrasound — Airway ultrasound is a non-invasive imaging allowing visualization and measurements of the tongue base and retrovascular fatty infiltration. Its main interest remains the evaluation of the tongue base which is clinically difficult.

SUMMARY:
Sleep apnea-hypopnea syndrome (SAHS) is a disorder of nocturnal ventilation due to the occurrence abnormally frequent pauses in breathing. It is a public health problem that currently affects 13 % of men and 6% of women between 30 and 70 years old. Sleep apneas are conventionally divided into obstructive and central apneas, depending on the persistence or no respiratory movements and the existence or not pharyngeal collapse during apnea. There are upper airway characterization studies (VAS) in patients with syndrome sleep apnea/hypopnea (OSAS). These physiological characterization studies (measurement of critical closing pressure (Pcrit) of the VAS) and anatomical (transcutaneous ultrasound of the muscles of the floor of the mouth, the base of the tongue, or by a acoustic pharyngometry of the VAS) are interested separately to different parameters without searching correlation with the severity of sleep apnea nor their potential as a screening tool for OSAS in patients at risk. The investigators hypothesize that a strong correlation and constant exists between the physiological collapsibility of VAS, the anatomical measurements of the VAS and the degree of severity of OSAS. Thus, the aim of this descriptive study is to characterization as complete as possible of the VAS of apneic patients in a homogeneous population and a better understanding of the pathophysiological obstructive events in patients without factor obvious risk.

DETAILED DESCRIPTION:
Obstructive sleep apnea-hypopnea syndrome (OSAS) is a nocturnal respiratory disorder caused by a succession of respiratory pauses. The prevalence of OSAHS has increased over the past two decades partly due to the fact that it is more often diagnosed but also due to the progression of obesity. It now affects 13% of men and 6% of women between the ages of 30 and 70. Sleep apneas are conventionally divided into obstructive and central apneas, depending on whether or not respiratory movements persist and whether or not there is pharyngeal collapse during the apnea. Continuous positive airway pressure (CPAP) ventilation via a nasal or naso-buccal mask is the reference treatment. The effectiveness of CPAP is directly linked to its observance. A well conducted treatment allows a significant improvement of symptoms related to OSAHS and effectively reduces daytime sleepiness. In the longer term, it would provide protection against cardiovascular events.

The physiopathology of obstructive apnea has been the subject of in-depth studies; the most recent data show that it is a multifactorial disease. Among the factors implicated, the investigators can cite pharyngeal anomalies (anatomy and collapsibility), a significant ventilatory response ("high loop gain") in response to variations in partial pressure of CO2 (pCO2), a weak pharyngeal muscle response during sleep and a high wakefulness threshold. Each of them can be evaluated by different methods: anatomy by a standardized clinical examination and imaging techniques, some of which have not yet been the subject of anatomo-functional correlation studies (such as the ultrasound or acoustic pharyngometry); collapsibility by measuring the critical closure pressure (Pcrit) (pressure applied at which closure of the airways is observed); the ventilatory response by analysis of the SpO2 and PCO2 signals in the exhaled air (PETCO2) in calm ventilation and ventilatory slope of response to hypercapnia; pharyngeal electromyogram and polysomnographic analysis.

The respective importance of these factors seems to vary greatly from one individual to another, but their characterization would make it possible to propose new avenues of treatment targeting the "loop gain", the pharyngeal muscle tone or the arousal threshold, and d adapt these targets to each patient for a personalized treatment.

The investigators hypothesize that a correlation exists between the physiological collapsibility of the VAS, the anatomical measurements of the VAS and the degree of severity of OSAHS. The objectives of our study are to identify clinical and physiological phenotypes of apneic patients, with the prospect of screening tools, a better distribution of targeted diagnostic and therapeutic resources.

ELIGIBILITY:
Inclusion criteria: - Any patient, consulting the sleep department of the Bichat hospital for suspected sleep apnea syndrome

* Patient for whom an PSG are prescribed as part of care
* Age ≥18 years and ≤85 years Exclusion criteria: - Recent ENT surgery (less than 6 months)
* Pregnancy in progress (declared)
* Pulsed oxyhaemoglobin saturation < 88% at rest on awakening
* Allergy to ultrasound gel
* Patient with difficulties in understanding the French language
* Vulnerable patient (guardianship, curators)
* Lack of affiliation to a social security scheme
* Lack of information and collection of informed, written and signed consent
* Patient under AME

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
measure of the values of critical closing pressure of the upper airway | during procedure
The measurements in cm of tissus thickness of the upper airways by ultrasound | during procedure
measure the cross-sectional area of the upper airway by a acoustic pharyngometry | during procedure

SECONDARY OUTCOMES:
measure of pharyngeal volume by ultrasound | during procedure
measure of pharyngeal collapsibility by ultrasound | during procedure
predictive value (Sp, Se) of acoustic pharyngometry measurements | during procedure
predictive value of ultrasound measurements (Sp, Se) | during procedure
measure of apnea hypopnea index by polysomnography | during procedure

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pia d'Ortho, MD. Ph.D, Principal Investigator — Assistance Publique - Hôpitaux de Paris (AP-HP)
Locations (1):
- Hôpital Bichat-Claude Bernard, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided